CLINICAL TRIAL: NCT07012538
Title: Renin-angiotensin System Inhibitor for Preventing Postoperative Recurrence of Stage II/III Colon Cancer
Brief Title: RASi for Preventing Postoperative Recurrence of Stage II/III Colon Cancer
Acronym: RAIPC
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Zhongshan Hospital Fudan University, Fudan University
Other Study IDs: RAIPC
Record Dates: First submitted 2025-05-30; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Colon Cancer (Stage II &Amp;Amp; III)
Keywords: renin-angiotensin system inhibitor; colon cancer; disease-free survival
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Renin-angiotensin system inhibitors (RASi): Using RASi after radical resection of stage II/III colon cancer
  Interventions: Drug: Renin-angiotensin system inhibitors (RASi)
- No renin-angiotensin system inhibitors (No RASi): Not using RASi after radical resection of stage II/III colon cancer
  Interventions: Drug: No renin-angiotensin system inhibitors (No RASi)

INTERVENTIONS:
Drug: Renin-angiotensin system inhibitors (RASi) — Using RASi after radical resection of stage II/III colon cancer for at least 3 years or till recurrence or death or inappropriate use of RASi.
  Groups: Renin-angiotensin system inhibitors (RASi)
Drug: No renin-angiotensin system inhibitors (No RASi) — Not using RASi after radical resection of stage II/III colon cancer for at least 3 years or till recurrence or death or needing RASi.
  Groups: No renin-angiotensin system inhibitors (No RASi)

SUMMARY:
The goal of this retrospective cohort study is to learn about the long-term effects of renin-angiotensin system inhibitors (RASi) in preventing patients with hypertension and stage II/III colon cancer from recurrence and metastases after radical resection. The main question it aims to answer is:

Does RASi improve the 3-year disease-free survival of patients with hypertension and stage II/III colon cancer after surgery? Participants with hypertension and already having radical resection of stage II/III colon cancer will be followed up for 3 years.

DETAILED DESCRIPTION:
Previous studies have shown that renin-angiotensin system inhibitors (RASi) may reduce postoperative recurrence and metastases of colorectal cancer. However, the relevant clinical evidences were low level and controversial. This study retrospectively collect patients with hypertension and stage II/III colon cancer after radical resection, and compare the patients with vs. without RASi in terms of long-term oncological outcomes, to study the inhibitory effect of RASi on recurrence and metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Inferior tumor edge > 15 cm from anal verge;
2. Received radical resection of primary tumor;
3. Pathological proved stage II or stage III adenocarcinoma;
4. No evidence of distant metastases at time of surgery (including pelvis, peritoneum, liver, lung, brain, bone, distant lymph node, etc), according to ultrasound, CT, MRI, PET-CT, intraoperative exploration, etc;
5. Combined with hypertension at time of surgery;
6. No other malignancies in medical history except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri;
7. Informed consent.

Exclusion Criteria:

1. Emergency surgery for acute intestinal obstruction, bleeding, perforation, etc;
2. Multiple primary colorectal cancer;
3. Hereditary colorectal cancer (familial adenomatosis polyposis, Lynch Syndrome, etc.);
4. Co-existent inflammatory bowel disease;
5. Pregnancy or lactation;
6. Received any of preoperative anti-cancer treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension and stage II/III colon cancer, received radical resection of the primary tumor.
Sampling Method: Non-Probability Sample
Enrollment: 2640 (Actual)
Dates: Start 2012-01-04 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years after surgery
  The events of 3-year disease-free survival are defined as any recurrence of metastases or death within 3 years after surgery.

OTHER OUTCOMES:
3-year overall survival | 3 years after surgery
  The events of 3-year overall survival are defined as any death within 3 years after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Whether to share the IPD will be decided after the research paper is published.